CLINICAL TRIAL: NCT04792060
Title: Prospective Study of the Management of Distal Ulna Fractures Using Hook Plate in Adult
Brief Title: Management of Distal Ulna Fractures Using Hook Plate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Fathy Tawfik, Resident, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-02-10
Record Dates: First submitted 2021-02-20; First posted 2021-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Distal Ulna Fractures
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adult patients with distal ulna fractures (Experimental): adult patients with distal ulna fractures
  Interventions: Procedure: Hook plate

INTERVENTIONS:
Procedure: Hook plate — We used titanium 2.4 mm hooked distal ulnar locked plate used for fixation of distal ulna fractures , this plate have low profile which is anatomically precontoured
  Other Names: Distal ulna anatomical plate

SUMMARY:
The aim of this current prospective study is to evaluate the effectiveness of an open reduction and internal fixation {ORIF} by distal ulna hooked locking compression plate (lcp) in treatment of isolated displaced distal ulna fracture in adult " without concomitant distal radius fractures.

DETAILED DESCRIPTION:
The distal ulna is an important component in the forearm and wrist motion. Pronation-supination is a complex movement, combining the rotation of the radius around the ulna with a horizontal and axial translation. If the distal ulna fails to heal in the proper anatomical position maintaining its original length with significant residual angulation at the fracture site, and separation of the DRUJ in a transverse axis, then a more severe limitation of forearm motion

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature distal ulna fracture with or without radius fracture.

Exclusion Criteria:

* Pathological fracture Skeletally immaturity Neurovascular problems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Management of Distal Ulna Fractures Using Hook Plate | 6 months
  surgery

CONTACTS AND LOCATIONS:
Overall Officials: salah roshdy ahmed, professor, Study Chair — Sohag University
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
• Patient still for 24 hours postoperative till discharge during this period follow up swelling and neurovascular complication and broad spectrum antibiotics will be taken.
  Follow up of cases at 2weeks postoperative 1-3-6 months.